CLINICAL TRIAL: NCT04263233
Title: Evaluation of the Optimal Transition Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH124_Optional Transition
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: ESRD; Hemodialysis
Keywords: ESRD; Hemodialysis; Education; Evaluation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Surveys and Questionnaires; Costs and Cost Analysis; Length of Stay

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Other: This program, which is provided for all patients new to dialysis at the participating units, will be evaluated by assessing patient clinical outcomes and the results of surveys measuring patient-reported symptoms, quality of life, knowledge and activation. In addition, satisfaction with the program will be assessed.
  Interventions: Other: Analysis using descriptive statistics of patient clinical outcomes.; Other: Surveys with participants using validated survey tools.; Other: Evaluation of the program process including time, costs, referral rates, admission to the program and length of stay.

INTERVENTIONS:
Other: Analysis using descriptive statistics of patient clinical outcomes. — Evaluation of the following:
  * Laboratory values at admission, week 4, and day 90.
  * Pre and post blood pressure at week one and week 4.
  * Intradialytic hypotension at week one and week 4.
  * Ultrafiltration rates at week one, week 4, day 90, day 180, and day 360.
  * Target weight defined and achievement in week one and week 4 and changes between week one and week 4.
  * Dialysis access type at week one and day 90.
  * Hospitalization and mortality rates.
Other: Surveys with participants using validated survey tools. — Surveys will assess participants' Symptom index, Quality of Life, Patient Activation as well as satisfaction with the program.
Other: Evaluation of the program process including time, costs, referral rates, admission to the program and length of stay. — Data will be collected using tracking tools throughout the program.

SUMMARY:
This is an evaluation of a program developed by a team of nephrologists, operations experts and researchers. The goal is to provide CKD patients with a better way to transition to life on dialysis - one that emphasizes even more individual clinical, psychosocial and lifestyle needs. On top of high-quality clinical care, the 4-week Optimal Transition program supports patients as they adjust to treatment and learn to live the best life possible. This is done through a robust education curriculum and a trust-building approach.

DETAILED DESCRIPTION:
In this program evaluation the investigators will be reporting on the following program outcomes:

1. Clinical and psychosocial stabilization: to include lab values, clinical dialysis parameters, patient-reported symptoms, quality of life, hospitalization and mortality rates.
2. Dialysis modality choice with satisfaction with the modality education and continued modality use over 24 months.
3. Patient knowledge, activation, and satisfaction.
4. Program parameters such as time, costs, referral rate, admissions and length of stay within the program.

ELIGIBILITY:
Inclusion Criteria:

* Referred for incenter hemodialysis at one of two Satellite Healthcare (SHC) participating dialysis units
* Without significant cognitive impairment;
* Able to meaningfully interact with staff; and
* Fluent in English (due to education material being limited to English at this time).

Exclusion Criteria:

* Unable to meaningfully interact with staff;
* Unable to read and understand English; or
* Has significant cognitive impairment per the nephrologist or Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred by their treating nephrologist to one of the two Satellite Healthcare (SHC) participating centers who are new to dialysis and meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-07-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical stabilization through standard clinical dialysis labs | On admission, week 4 and day 90
  Evaluation of changes in the Standard of care monthly dialysis labs
Evaluation of clinical stabilization through standard clinical dialysis blood pressure measurements | At week one and week 4.
  Evaluation of any changes in the Pre and post dialysis blood pressures for each patient which are collected as part of the patient's dialysis flow sheet.
Evaluation of clinical stabilization through standard clinical dialysis measurements of Intradialytic blood pressures | At week one and week 4.
  Evaluation of any changes in the incidence of Intradialytic hypotension as assessed by review of the patient's dialysis flow sheet.
Evaluation of clinical stabilization through standard clinical dialysis measurements of ultrafiltration | At week one, week 4, day 90, day 180 and day 360.
  Evaluation of interval changes in the patient's ultrafiltration rates as measured by the dialysis machine and reported on the patient's dialysis flow sheets.
Evaluation of clinical stabilization through standard clinical dialysis measurements of weight | At week one and week 4, and changes between week one and week 4.
  Target weight defined and achieved as measured by standard of care at the unit
Evaluation of clinical stabilization through standard clinical dialysis measurements | At week one and day 90
  Dialysis access type as reported in the dialysis treatment sheets
Evaluation of clinical stabilization through standard clinical dialysis collection of patient hospitalizations. | Day 30, day 90, 6 months and 12 months
  Hospitalization rates as reported in the standard dialysis record for all patients
Evaluation of clinical stabilization through standard clinical dialysis records. | Day 30, day 90, 6 months and 12 months
  Mortality rates as reported in the standard dialysis record for all patients
Evaluation of clinical and psychological stabilization through a quality of life measurement. | Week 4
  The EQ-5D tool will be used
Evaluation of clinical and psychological stabilization through assessment of patient symptoms. | Week 1 and Week 4
  The ESAS-r:Renal tool will be used
Satisfaction with the modality options education | Week 1 and Week 4
  Survey of patient experience
Type of Dialysis Modality chosen by the patient | Week 1 and Week 4
  Dialysis modality choice as reported by the patient
Actual Type of Dialysis Modality used by the patient | week 4, month 3, 6, 12, 18 and 24
  Dialysis modality as reported on the standard dialysis treatment sheets
Evaluation of patient knowledge of dialysis and modalities | Week 1, 2, 3, 4
  Weekly focused one on one discussion where the patient is questioned about his/her understanding of dialysis, his/her progress, questions, concerns using a questionnaire developed by the investigator
Evaluation of patient activation | Week 3 and month 3
  Survey measuring patient activation (PAM-13) survey
Evaluation of patient satisfaction | Week 4 or discharge from the program whichever comes first
  Survey of satisfaction with the program
Evaluation of the program process for time utilization | Week 1 through week 4
  Time per patient for visits from program start to completion for each patient
Evaluation of the program process for cost utilization | Week 1 through week 4
  Time, and thus cost, for personnel to complete the program with each patient from entrance to completion or early termination.
Evaluation of the feasibility of the program | Week 1 through week 4
  Number of referrals to the program and subsequent number of admissions to the program.
Evaluation of the program efficiency | Week 1 through week 4
  Average length of stay for each patient in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Hussein, MBBS, Principal Investigator — Satellite Healthcare, Inc.
Locations (3):
- United States (3):
  - Satellite Healthcare Oakland, Oakland, California
  - Satellite Healthcare Sacramento, Sacramento, California
  - Satellite Healthcare Chickasaw Gardens, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No